CLINICAL TRIAL: NCT01707706
Title: A Randomized Controlled Trial of Electroacupuncture for Persistent Insomnia Symptoms Associated With Major Depressive Disorder
Brief Title: Acupuncture for Persistent Insomnia Associated With Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACUP-004
Record Dates: First submitted 2012-02-22; First posted 2012-10-16 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Insomnia; Depression
Keywords: Insomnia; Depression; Electroacupuncture; Acupuncture; Randomized Clinical Trial; Traditional Chinese Medicine
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression | interventions — Acupuncture Therapy; Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Traditional Acupuncture (Experimental): Patients will be treated at bilateral Ear Shenmen, Sishencong EX-HN1, Anmian, Neiguan PC6, Shenmen HT7, Sanyinjiao SP6, and unilateral Yintang EX-HN3 and Baihui GV20. Acupuncture treatment will be performed by a registered Chinese medicine practitioner. "De qi"(an irradiating feeling considered to be indicative of effective needling) is achieved if possible. An electric-stimulator (ITO ES160, Japan) is connected to these needles to give an electric-stimulation in continuous wave, frequency of 4 Hz, 0.4 ms square wave pulses and constant current. Surgical tape or hair pin will be adhered to the needles.The needles will be left for 30 min and then removed. Acupuncture treatment will consist of three sessions per week for 3 consecutive weeks.
  Interventions: Other: Acupuncture
- Minimal Acupuncture (Active Comparator): Patients will be treated superficially at points away from classic acupoints. The points include bilateral "Forearm" [1 inch lateral to the middle point between HE3 and HE7] , "Upper arm" [1 inch lateral to LU 3 ], and "Lower leg" [0.5 inch dorsal to GB39]; for head, the non-acupoints include bilateral "Head" [middle point between GB8 and ST8], "Forehead" [middle point between ST8 and GB14], "Neck" [middle point between TB16 and SI17], and "Ear" [the point on the helix, inferior to the apex]. The points selected have been used in previous acupuncture studies as sham control. "De qi" is avoided during needling. The treatment procedure, electric-stimulation, frequency, duration and number of treatment sessions will be the same for the Traditional Acupuncture group.
  Interventions: Other: Acupuncture
- Placebo Acupuncture (Placebo Comparator): Placebo needles designed by Streitberger (1998) will be used. The placebo needles are blunt needle that will not penetrate the skin during needle insertion. The handles of these placebo needles will slide over the needle when it is compressed, giving it the appearance of penetrating the skin. The placebo needles are inserted to the site 1 inch beside the acupoints in order to avoid the acupressure effect. The needles are held by a surgical tape or hair pin in hairy region to imitate the retention of needles. The needles are connected to an electric-stimulator with zero frequency and amplitude. The number, duration and frequency of the treatment sessions, and the intervention procedure will be the same for electro-acupuncture and placebo acupuncture.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture at bilateral Ear Shenmen, Sishencong EX-HN1 , Anmian , Neiguan PC6 , Shenmen HT7 , Sanyinjiao SP6 , and unilateral Yintang EX-HN3 and Baihui GV20. The needles will be left for 30 min and then removed. Acupuncture treatment will consist of three sessions per week for 3 consecutive weeks.
  Other Names: Electroacupuncture

SUMMARY:
The purpose of this study is to evaluate the clinical effectiveness of acupuncture treatment on residual insomnia in major depressive patients.

DETAILED DESCRIPTION:
This is a randomized single-blinded controlled trial. Patients will be randomly assigned to one of the three groups. One is the traditional acupuncture treatment group, one is the non-traditional acupuncture treatment group and the other is an acupuncture-like placebo treatment. Patients will be put into groups and then compared. The chance of getting into each group is 2:2:1.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above
* A previous Diagnostic and Statistical Manual of Mental Disorders-IV Major Depressive Disorder
* Have a current Diagnostic and Statistical Manual of Mental Disorders-IV diagnosis of insomnia disorder
* Insomnia more than 3 nights per week for at least 3 months
* Insomnia Severity Scale (ISI) total score higher than 15 at screening and baseline visit
* Use of antidepressants at the same dosage for at least 12 weeks prior to screening visit
* Hypnotic dosage has not been increased in the last 4 weeks

Exclusion Criteria:

* Have a Hamilton Depression Rating Scale scores above 18
* Have sleep apnea or periodic limbs movement disorder detected by overnight polysomnography
* Have suicidal risk as assessed by the Hamilton Depression Rating Scale suicidal risk item
* Have previous history of schizophrenia, other psychotic disorders, and bipolar disorder
* Have current alcohol or drug abuse and dependence
* Pregnant, breast-feeding, or woman of childbearing potential not using adequate contraception
* Have infection or abscess close to the site of selected acupoints and in the investigator's opinion inclusion is unsafe
* Taking Chinese herbal medicine or over-the-counter drugs which are intending for insomnia within the last 2 weeks prior to baseline or during the study
* Any acupuncture treatment during the previous 12 months prior to baseline and
* Unstable medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Self-rated sleep quality score changes from baseline to 5-week posttreatment measured by Insomnia Severity Index questionnaire | Baseline, 1-week and 5-week posttreatment.

SECONDARY OUTCOMES:
Self-rated sleep quality score measured by the Pittsburgh Sleep Quality Index (PSQI) questionnaire | Baseline, 1-week posttreatment, and 5-week posttreatment.
Depression state measured by Hamilton Depression Rating Scale (HAMD) | Baseline, 1-week posttreatment, and 5-week posttreatment.
Depression state measured by Hamilton Anxiety Rating Scale (HAMA) | Baseline, 1-week posttreatment, and 5-week posttreatment
Subjective report of painful and non-painful somatic symptoms measured by Somatic Symptom Inventory (SSI) | Baseline, 1-week posttreatment, and 5-week posttreatment.
Subjects' functioning regarding work/study, social life and family measured by Sheehan Disability Scale (SDS) | Baseline, 1-week posttreatment and 5-week posttreatment
Self-rated severity of depressive and anxiety symptoms measured by Hospital Anxiety and Depression Scale (HADS) | Baseline, 1-week posttreatment, and 5-week posttreatment
Self-rated assessment regarding the degree of catastrophic thoughts about pain measured by Pain Catastrophizing Scale (PCS) | Baseline, 1-week posttreatment, and 5-week posttreatment.
Subjects' general health and quality of life regarding physical functioning, social functioning, physical role limitations, emotional role limitations, mental health, vitality, bodily pain, and general health perception measured by Short form -36 (SF-36) | Baseline, 1-week posttreatment, and 5-week posttreatment.
Self-rated fatigue score measured by Multidimensional Fatigue Inventory (MFI) | Baseline, 1-week posttreatment, and 5-week posttreatment
Subjects' credibility to the treatment measured by Credibility of treatment rating scale | Baseline, second treatment (expected 3-day post-baseline ) and the last time of the treatment (expected 19-day post-baseline )
Serious adverse events measured by Serious Adverse Event (SAE) | 1-week, 2-week, and 3-week post-baseline, 1-week and 5-week posttreatment
Potential adverse events related to acupuncture measured by Adverse Events Report Related to Acupuncture | 1-week, 2-week, and 3-week post-baseline, 1-week and 5-week posttreatment
Sleep parameters (sleep onset latency, sleep efficiency, total sleep time, times of wakening during sleep) changes from baseline to 5-week posttreatment by objective measure - wrist actigraphy | Baseline, 1-week posttreatment, and 5-week posttreatment.
Sleep parameters (sleep onset latency, sleep efficiency, total sleep time, times of wakening during sleep) changes from baseline to 5-week posttreatment by subjective measures using sleep log. | Baseline, 1-week posttreatment, and 5-week posttreatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Fai Chung, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Western Psychiatry Centre, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Yeung WF, Chung KF, Yu YB, Lao L. What predicts a positive response to acupuncture? A secondary analysis of three randomised controlled trials of insomnia. Acupunct Med. 2017 Mar;35(1):24-29. doi: 10.1136/acupmed-2016-011058. Epub 2016 Aug 8. PMID 27503746
- [Derived] Yeung WF, Chung KF, Yu BY, Lao L. Response to placebo acupuncture in insomnia: a secondary analysis of three randomized controlled trials. Sleep Med. 2015 Nov;16(11):1372-1376. doi: 10.1016/j.sleep.2015.07.027. Epub 2015 Aug 31. PMID 26498238
- [Derived] Chung KF, Yeung WF, Yu YM, Yung KP, Zhang SP, Zhang ZJ, Wong MT, Lee WK, Chan LW. Acupuncture for residual insomnia associated with major depressive disorder: a placebo- and sham-controlled, subject- and assessor-blind, randomized trial. J Clin Psychiatry. 2015 Jun;76(6):e752-60. doi: 10.4088/JCP.14m09124. PMID 26132682
- [Derived] Chung KF, Yeung WF, Kwok CW, Yu YM. Risk factors associated with adverse events of acupuncture: a prospective study. Acupunct Med. 2014 Dec;32(6):455-62. doi: 10.1136/acupmed-2014-010635. Epub 2014 Sep 30. PMID 25271149